CLINICAL TRIAL: NCT06394102
Title: Visual Health Evaluation of Natural Color Display Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: TREC2023-KY120
Record Dates: First submitted 2024-04-08; First posted 2024-05-01 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-03

CONDITIONS: Chromatic Adaptation
Keywords: Chromatic adaptation; Reading efficiency; Visual function; Visual fatigue; Fundus blood flow
MeSH Terms: conditions — Asthenopia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Group (Experimental): Is a group that accepts natural color mode processing and then accepts natural color mode closing. In this group, subjects will first be exposed to an environment using a natural color pattern, which applies a specific light source to adjust the color temperature of the ambient light, and the phone color temperature will change with the ambient light color temperature. To evaluate the effects of natural color patterns on visual fatigue and visual function, including but not limited to measures of adjustment function, assembly function, reading efficiency, blink detection, and retinal fundus blood flow.
  Interventions: Other: The automatic color temperature adjustment mode equipped on terminal display devices can reduce the discrepancy between the color temperature of the device and the ambient light.
- B Group (Experimental): Is the group that accepts the natural color mode off first, and then accepts the natural color mode on. In group B, the subjects will first be in the condition of changing ambient light, and the color temperature of the phone will not change with the ambient light color temperature. Then the experiment was performed on different days to open the natural color mode. The aim is to provide a benchmark against which to compare the effects of natural color pattern treatment in the experimental group.
  Interventions: Other: The automatic color temperature adjustment mode equipped on terminal display devices can reduce the discrepancy between the color temperature of the device and the ambient light.

INTERVENTIONS:
Other: The automatic color temperature adjustment mode equipped on terminal display devices can reduce the discrepancy between the color temperature of the device and the ambient light. — A program mode on a terminal display device that reduces the difference between the color temperature of the ambient light and that of the display device.
  Other Names: Automatic color temperature adjustment mode equipped on terminal display devices.

SUMMARY:
Study on visual fatigue and visual function under changing ambient light color temperature by natural color mode: The influence of electronic display devices on visual fatigue of human eyes is the main evaluation index and the main outcome index of this experiment. Secondary outcome indicators were visual function indicators such as regulation and aggregation. There are other outcome measures: effective reading efficiency, blink detection, retinal fundus blood flow. The baseline values of the above indicators were respectively measured, and then the specific values of different indicators when the natural color mode was enabled and not enabled were collected under the changing ambient light color temperature, and the baseline values were statistically compared and analyzed. Evaluate the effect of natural color patterns on the relief of visual fatigue and on visual function.

ELIGIBILITY:
Inclusion Criteria:

1. Adult population, regardless of gender
2. Refractive error is less than or equal to -2.5D and both eyes achieve corrected visual acuity of 0.8 or higher.
3. Normal intraocular pressure with no organic pathology.
4. No apparent symptoms of dry eye.
5. Willing to cooperate to complete all the tests.
6. Voluntarily signing the informed consent form.

Exclusion Criteria:

* 1: Individuals with strabismus and amblyopia exist.

  2: Suffering from congenital eye conditions such as congenital cataracts or congenital retinal diseases.

  3: Those who have undergone intraocular surgery (such as cataract removal, intraocular lens implantation, etc.).

  4: Individuals with refractive media opacity (such as corneal lesions, lens opacity, etc.).

  5: Abnormal intraocular pressure (IOP) (IOP < 10 mmHg or IOP > 21 mmHg, or a bilateral IOP difference of ≥5 mmHg).

  6: Only one eye meets the inclusion criteria.

  7: Active corneal infections such as bacterial, fungal, viral, or other acute or chronic anterior segment inflammations.

  8: Currently using medications that may lead to dry eye or affect vision and corneal curvature.

  9: Other ocular conditions, such as dacryocystitis, eyelid disorders and abnormalities, abnormal intraocular pressure, and glaucoma.

  10: Unable to undergo regular eye examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Visual fatigue | Each participant will complete the visual fatigue questionnaire, followed immediately by a VEP task, and then re-assess visual fatigue immediately afterward. This sequence will occur twice per group, totaling four assessments per participant.
  The visual fatigue questionnaire utilized in this study consists of a self-report survey with a total of 19 items. It is designed to comprehensively assess the severity of visual fatigue symptoms, with a scoring system ranging from 1 to 7. Higher scores indicate more severe symptoms, encompassing three primary domains: ocular symptoms, visual discomfort, and psychological aspects triggered by visual fatigue.

SECONDARY OUTCOMES:
Measurement of Accommodative Sensitivity with Flip-Chart Post-VEP Tasks | Each participant will have three measurements: a baseline, and two post-VEP tasks, with immediate flip-chart tests after each task.
  This clinical study involves the assessment of accommodative sensitivity for both monocular and binocular vision using a flip-chart immediately following each visual evoked potential (VEP) task. The measurement will quantify the number of optotypes correctly identified within one minute, indicative of the subject's accommodative capacity.
AC/A Ratio Measurement Post-VEP Tasks | Each participant will undergo three AC/A ratio measurements: at baseline and immediately after each of two VEP tasks.
  This study involves the measurement of the AC/A ratio, which is a critical parameter in binocular vision assessment, reflecting the relationship between accommodation (focus adjustment) and convergence (ocular alignment). The AC/A ratio will be determined using the prism bar technique, which involve adding lenses to stimulate accommodation and measuring the resulting changes in convergence.
Ocular Fundus Blood Flow | Retinal blood flow measurements should be taken within 3 minutes after the completion of each visual evoked potential (VEP) task. There are two VEP tasks per group, along with a baseline measurement, resulting in a total of three measurements.
  The study measured the sub foveal choroidal thickness, superficial vessel complex (SVC) density, and deep vessel complex (DVC) density, analyzing changes in retinal blood flow under the two modes.
Blink Frequency | Blink frequency 3 minutes after the start of each visual evoked task and 3 minutes before the end
  Use electronic devices to record the number of clicks within 3 minutes and calculate the frequency.
Reading efficiency | The test was recorded 10 minutes after the start and 10 minutes before the end.
  The number pairs were read in the first and last 10 minutes of the visual evoked task, and the number of number pairs read per minute was counted.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospitol,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No